CLINICAL TRIAL: NCT03735784
Title: Brief Group MI Intervention for AOD Use and Sexual Risk Behavior in Homeless Youth
Brief Title: Intervention for Substance Use and Sexual Risk Behavior in Homeless Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Joan Tucker, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01AA025641 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Substance Use; Unprotected Sex
MeSH Terms: conditions — Substance-Related Disorders; Unsafe Sex

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWARE condition (Experimental): AWARE is a four-session Motivational Interviewing (MI)-informed group risk reduction intervention that incorporates education, skills building and personalized feedback.
  Interventions: Behavioral: AWARE
- Standard Care condition (No Intervention): Participants in the Standard Care condition have access to "usual care" at the drop-in center where the study is being conducted.

INTERVENTIONS:
Behavioral: AWARE — AWARE consists of four group sessions. The AWARE curriculum involves sharing basic information on sexually transmitted diseases; providing condom use skills training; providing normative feedback on substance use and sexual risk behavior among young adults; discussing unrealistic beliefs about substance use and sexual risk; discussing potential benefits of both cutting down and stopping risky behaviors; and discussing risky situations and coping strategies.
  Arms: AWARE condition

SUMMARY:
This study will evaluate a program called AWARE, which is a voluntary four session group-based motivational interviewing (MI) intervention to reduce substance use and sexual risk behavior among 18-25 year olds who are experiencing homelessness. The hypothesis is that participants who receive AWARE will show greater reductions in substance use and sexual risk behavior over a 12 month period compared to participants who do not receive the program.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 25; seeking services at one of the participating drop-in centers; no cognitive impairment observed during the screening process; planning to be in the study area for the next month; has either an email account or cell phone where they can be reached; and English speaking.

Exclusion Criteria:

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Substance use | 12 months
  frequency and quantity of alcohol and drug use
Unprotected sex | 12 months
  proportion of condom-unprotected sexual events

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - My Friend's Place, Hollywood, California
  - Youth Center on Highland, Los Angeles, California
  - Safe Place for Youth, Venice Beach, California

REFERENCES:
- [Derived] DiGuiseppi G, Jose R, D'Amico EJ, Klein DJ, Rodriguez A, Pedersen ER, Tucker JS. Investigating Change in Psychosocial Outcomes for Young Adults Experiencing Homelessness in Los Angeles With and Without Pregnancy Experiences. Perspect Sex Reprod Health. 2025 Sep;57(3):329-339. doi: 10.1111/psrh.70028. Epub 2025 Jul 29. PMID 40728251
- [Derived] DiGuiseppi G, Pedersen ER, Brown ME, Rodriguez A, Jose R, Klein DJ, D'Amico EJ, Tucker JS. Protective behavioral strategies and alcohol consequences following a group-based motivational intervention for young adults experiencing homelessness. Psychol Addict Behav. 2025 Sep;39(6):516-527. doi: 10.1037/adb0001047. Epub 2025 Jan 9. PMID 39786835
- [Derived] Tucker JS, D'Amico EJ, Rodriguez A, Garvey R, Pedersen ER, Klein DJ. A randomized controlled trial of a brief motivational interviewing-based group intervention for emerging adults experiencing homelessness: 12-Month effects on substance use and sexual risk behavior. J Subst Use Addict Treat. 2023 Sep;152:209114. doi: 10.1016/j.josat.2023.209114. Epub 2023 Jun 22. PMID 37355155
- [Derived] Tucker JS, D'Amico EJ, Pedersen ER, Rodriguez A, Garvey R. Study protocol for a group-based motivational interviewing brief intervention to reduce substance use and sexual risk behavior among young adults experiencing homelessness. Addict Sci Clin Pract. 2020 Jul 28;15(1):26. doi: 10.1186/s13722-020-00201-x. PMID 32723349